CLINICAL TRIAL: NCT05449431
Title: Comparison of the 1-min Sit-to-Stand Test to the 6-minute Walk Test in the Respiratory Functional Assessment of Pulmonary Fibrosis: a Cross-over Trial
Brief Title: Comparison of the 1-min Sit-to-Stand Test to the 6-minute Walk Test in the Respiratory Functional Assessment of Pulmonary Fibrosis
Acronym: LaMinute_FIP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: LaMinute_FIP
Record Dates: First submitted 2022-06-29; First posted 2022-07-08 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TLC1_TM6 (Experimental): Patient doing 1-minute chair lift test (TLC1) before 6-minute Walk Test (TM6).
  Interventions: Other: TLC1_TM6
- TM6_TLC1 (Experimental): Patient performing 6-minute Walk Test (TM6) before 1-minute chair lift test (TLC1)
  Interventions: Other: TM6_TLC1

INTERVENTIONS:
Other: TLC1_TM6 — Following this inclusion, patients are performing 1-minute chair lift test (TLC1) before 6-minute Walk Test (TM6). Each exercise will be separated by 30 minutes during which the patient will be sitting in a waiting room.
  Arms: TLC1_TM6
Other: TM6_TLC1 — Following this inclusion, patients are performing 6-minute Walk Test (TM6) before 1-minute chair lift test (TLC1). Each exercise will be separated by 30 minutes during which the patient will be sitting in a waiting room.
  Arms: TM6_TLC1

SUMMARY:
Fibrosing interstitial lung diseases or pulmonary fibrosis represent a heterogeneous group of progressive pulmonary pathologies, responsible for a significant morbi-mortality. They are defined by an infiltration of the pulmonary interstitium associating in a variable way an inflammatory component (deposit of inflammatory cells) and a fibrosing component (deposit of collagen). Idiopathic pulmonary fibrosis (IPF) is the most common and most severe pulmonary fibrosis. Other pulmonary fibroses are mainly represented by non-specific interstitial lung disease, pulmonary fibroses associated with connectivites, hypersensitivity pneumonitis, certain pneumoconiosis (occupational diseases) and sarcoidosis. The process of fibrosis is responsible for a loss of elasticity of the lung, leading to a decrease in lung volumes associated with an alteration of gas exchange.

In these diseases, the clinician must be able to rely on reliable means to assess the severity of the disease based mainly on the measurement of lung volumes and gas exchange, at diagnosis and in the follow-up of the patient, in order to propose the most appropriate management. Lung volumes are assessed by respiratory function tests. Forced vital capacity is the reference volume value used. Impaired gas exchange is assessed at rest by measuring carbon monoxide diffusion capacity, arterial oxygen saturation and arterial blood gases.

The functional capacity to exercise is also a very important evaluation criterion in terms of prognosis and in the follow-up of the patient. It is assessed by means of ergocycle tests which mainly determine the maximal oxygen consumption. These are relatively complex tests that require special equipment and are not routinely performed. Simpler field tests have been developed to assess functional capacity during exercise, the most widely used and validated being the 6-minute Walk Test (TM6).

Other field tests to assess functional capacity to exercise have been developed, such as the 30-second, 1-minute, and 3-minute chair lift tests, stepper tests, and step and stair tests. Among them, the 1-minute chair lift test (TLC1) is the best evaluated. It consists of sitting down and getting up from a chair as many times as possible in 1 minute. The criteria measured are mainly the number of lifts and desaturation. Thus, the fundamental advantage of the TLC1 over the TM6 is the exemption from temporal and spatial constraints since it takes only a few minutes and can be performed in a medical office. While TLC1 seems to be the most suitable, there are still a few pitfalls in substituting TLC1 for TM6 during diffuse interstitial lung disease.

First, there is only one study reporting the results of TLC1 in a healthy population. It provides a chart of results according to age. Unfortunately, only the number of lifts is reported without any data on heart rate, SaO2 or sensation of dyspnea.

In respiratory pathologies, TLC1 has been studied mainly in patients with chronic obstructive pulmonary disease (COPD) and little in PID. Unlike TM6, TLC1 is reproducible and has no learning effect in this population. Interestingly, one study found that peak desaturation and peak oxygen consumption occurred during the recovery phase some seconds after the end of the test.

Studies on TLC1 during SID do not allow us to conclude that this test can substitute for TM6. However, investigators may note certain limitations, in particular the small number of patients studied and the retrospective nature of the 2 largest of them. Above all, it seems that the use of TLC1 could be optimized by taking into account the recovery phase in the evaluation of desaturation.

The hypothesis of our study is that the TLC1 taking into account the recovery phase can replace the TM6 in the management of fibrosing PID for prognostic evaluation, patient follow-up and indication of oxygen therapy. It is more accessible and its use by all practitioners in face-to-face or telemedicine would allow a better management of these patients. Finally, the investigators hypothesize that the TLC1 will result in lower costs in the management of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age is ≥ 18 years
* Patient with fibrosing interstitial lung disease
* French-speaking patient
* Patient affiliated to a health insurance plan
* Patient who has given free, informed and written consent

Exclusion Criteria:

* Patient with an exacerbation of fibrosis in the last 6 months
* Patient with comorbidities limiting exercise performance
* Distance traveled < 200m at TM6
* Patient on long-term oxygen therapy (LTO)
* Patient already included in a type 1 interventional research protocol (RIPH1)
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under court protection
* Pregnant or breastfeeding patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-08-08 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-12-05 (Estimated)

PRIMARY OUTCOMES:
Strength of the relationship between O2 desaturation obtained with WT-6 and TLC1 at Day 1 | Day 1
  This outcome corresponds to the difference of O2 desaturation obtained with TM6 and TLC1.

SECONDARY OUTCOMES:
Equivalence of the percentage of desaturation on the TM6 and the TLC1 | Month 6
  This outcome corresponds to the Difference between initial SaO2 and final SaO2. The objective is to test the equivalence of the percentage of desaturation between these 2 parameters obtained with the TM6 and the TLC1.
Strength of the relationship between O2 desaturation obtained with WT-6 and TLC1 at month 6 | Month 6
  This outcome corresponds to nadir of O2 desaturation obtained with TM6 and TLC1.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Marc NACCACHE, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Background] Holland AE, Spruit MA, Troosters T, Puhan MA, Pepin V, Saey D, McCormack MC, Carlin BW, Sciurba FC, Pitta F, Wanger J, MacIntyre N, Kaminsky DA, Culver BH, Revill SM, Hernandes NA, Andrianopoulos V, Camillo CA, Mitchell KE, Lee AL, Hill CJ, Singh SJ. An official European Respiratory Society/American Thoracic Society technical standard: field walking tests in chronic respiratory disease. Eur Respir J. 2014 Dec;44(6):1428-46. doi: 10.1183/09031936.00150314. Epub 2014 Oct 30. PMID 25359355
- [Background] Nathan SD, du Bois RM, Albera C, Bradford WZ, Costabel U, Kartashov A, Noble PW, Sahn SA, Valeyre D, Weycker D, King TE Jr. Validation of test performance characteristics and minimal clinically important difference of the 6-minute walk test in patients with idiopathic pulmonary fibrosis. Respir Med. 2015 Jul;109(7):914-22. doi: 10.1016/j.rmed.2015.04.008. Epub 2015 Apr 24. PMID 25956020
- [Background] American Thoracic Society. Idiopathic pulmonary fibrosis: diagnosis and treatment. International consensus statement. American Thoracic Society (ATS), and the European Respiratory Society (ERS). Am J Respir Crit Care Med. 2000 Feb;161(2 Pt 1):646-64. doi: 10.1164/ajrccm.161.2.ats3-00. No abstract available. PMID 10673212
- [Background] Lama VN, Flaherty KR, Toews GB, Colby TV, Travis WD, Long Q, Murray S, Kazerooni EA, Gross BH, Lynch JP 3rd, Martinez FJ. Prognostic value of desaturation during a 6-minute walk test in idiopathic interstitial pneumonia. Am J Respir Crit Care Med. 2003 Nov 1;168(9):1084-90. doi: 10.1164/rccm.200302-219OC. Epub 2003 Aug 13. PMID 12917227
- [Background] AARC clinical practice guideline. Exercise testing for evaluation of hypoxemia and/or desaturation. American Association for Respiratory Care. Respir Care. 1992 Aug;37(8):907-12. No abstract available. PMID 10145783
- [Background] du Bois RM, Weycker D, Albera C, Bradford WZ, Costabel U, Kartashov A, Lancaster L, Noble PW, Sahn SA, Szwarcberg J, Thomeer M, Valeyre D, King TE Jr. Six-minute-walk test in idiopathic pulmonary fibrosis: test validation and minimal clinically important difference. Am J Respir Crit Care Med. 2011 May 1;183(9):1231-7. doi: 10.1164/rccm.201007-1179OC. Epub 2010 Dec 3. PMID 21131468
- [Background] Cottin V, Bonniaud P, Cadranel J, Crestani B, Jouneau S, Marchand-Adam S, Nunes H, Wemeau-Stervinou L, Bergot E, Blanchard E, Borie R, Bourdin A, Chenivesse C, Clement A, Gomez E, Gondouin A, Hirschi S, Lebargy F, Marquette CH, Montani D, Prevot G, Quetant S, Reynaud-Gaubert M, Salaun M, Sanchez O, Trumbic B, Berkani K, Brillet PY, Campana M, Chalabreysse L, Chatte G, Debieuvre D, Ferretti G, Fourrier JM, Just N, Kambouchner M, Legrand B, Le Guillou F, Lhuillier JP, Mehdaoui A, Naccache JM, Paganon C, Remy-Jardin M, Si-Mohamed S, Terrioux P; OrphaLung. [French practical guidelines for the diagnosis and management of IPF - 2021 update, short version]. Rev Mal Respir. 2022 Mar;39(3):275-312. doi: 10.1016/j.rmr.2022.01.005. Epub 2022 Mar 15. French. PMID 35304014
- [Background] Singh SJ, Puhan MA, Andrianopoulos V, Hernandes NA, Mitchell KE, Hill CJ, Lee AL, Camillo CA, Troosters T, Spruit MA, Carlin BW, Wanger J, Pepin V, Saey D, Pitta F, Kaminsky DA, McCormack MC, MacIntyre N, Culver BH, Sciurba FC, Revill SM, Delafosse V, Holland AE. An official systematic review of the European Respiratory Society/American Thoracic Society: measurement properties of field walking tests in chronic respiratory disease. Eur Respir J. 2014 Dec;44(6):1447-78. doi: 10.1183/09031936.00150414. Epub 2014 Oct 30. PMID 25359356
- [Background] Strassmann A, Steurer-Stey C, Lana KD, Zoller M, Turk AJ, Suter P, Puhan MA. Population-based reference values for the 1-min sit-to-stand test. Int J Public Health. 2013 Dec;58(6):949-53. doi: 10.1007/s00038-013-0504-z. Epub 2013 Aug 24. PMID 23974352
- [Background] Gephine S, Bergeron S, Tremblay Labrecque PF, Mucci P, Saey D, Maltais F. Cardiorespiratory Response during the 1-min Sit-to-Stand Test in Chronic Obstructive Pulmonary Disease. Med Sci Sports Exerc. 2020 Jul;52(7):1441-1448. doi: 10.1249/MSS.0000000000002276. PMID 31977637